CLINICAL TRIAL: NCT05003856
Title: Radiofrequency Ablation Use in Thyroid Nodule
Brief Title: Radiofrequency Ablation for the Treatment of Benign or Low Risk Thyroid Nodule
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrativley Complete, 75%<Participants
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0542; NCI-2021-08354 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0542 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-05; First posted 2021-08-12 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Benign Thyroid Gland Neoplasm; Recurrent Thyroid Gland Carcinoma; Thyroid Gland Follicular Tumor of Uncertain Malignant Potential; Thyroid Gland Nodule; Thyroid Gland Papillary Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule; Thyroid Cancer, Papillary | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (RFA) (Experimental): Patients undergo ultrasound guided RFA over 1-2 hours.
  Interventions: Other: Quality-of-Life Assessment; Procedure: Radiofrequency Ablation

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Radiofrequency Ablation — Undergo RFA
  Other Names: Ablation, Radiofrequency; Radiofrequency Interstitial Ablation; RFA

SUMMARY:
This phase IV trial studies the effect of radiofrequency ablation in treating patients with benign or low risk thyroid nodule. Radiofrequency ablation uses a needle to deliver a high-frequency electric current to kill tumor cells by heating them. The goal of this research study is to learn if ultrasound guided radiofrequency ablation can provide the same treatment result as standard surgical removal of the thyroid nodule, small primary thyroid, or thyroid cancers that have come back. Researchers also want to learn if the procedure can be less invasive and perhaps provide a better recovery response than surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the longitudinal thyroid nodule volume changes induced by radiofrequency ablation (RFA) during post procedure follow-up.

SECONDARY OBJECTIVES:

I. Evaluate treatment response to compressive and/or cosmetic symptoms that affect patient's quality of life.

II. Evaluate the sonographic features of the nodule induced by RFA.

III. Compare cost of ultrasound guided RFA to gold standard surgical thyroidectomy.

OUTLINE:

Patients undergo ultrasound guided RFA over 1-2 hours.

After completion of study treatment, patients are followed up at 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient is older than 18 years, is not a surgical candidate or refuses to have surgery
* Patient is medically fit to undergo local anesthesia with or without conscious sedation
* Patient is able to understand and give consent to participation in the study
* Presence of compression symptoms or cosmetic concerns for which patient request treatment of the benign thyroid nodule
* Solitary thyroid nodule or dominating nodule that is well-defined in multinodular goiter
* Benign nodule is >= 2 cm in the largest dimension, and has either solid, or predominantly solid composition (>= 70% volume) without large calcification. Nodule is confirmed as benign (Bethesda II) on at least 2 ultrasound guided fine needle aspirations (FNA) or core needle biopsy (CNB) or a single benign diagnosis of FNA or CNB when the nodule has benign ultrasound features (American College of Radiology [ACR] Thyroid Imaging Reporting & Data System [TI-RAD] TR 1-3, American Thyroid Association [ATA] very low suspicion) within 6 months of planned RFA
* Indeterminate thyroid nodule (atypical cells of undetermined significance [ACUS], follicular neoplasm), papillary thyroid carcinoma (PTC) without metastasis or locally recurrent thyroid cancer < 2 cm in the largest dimension. Nodule cytology is confirmed on a single FNA or CNB when the nodule has concordant ultrasound features (ACR TI-RAD TR 4-5, ATA intermediate-high suspicion) within 6 months of planned RFA
* Entirety of the selected nodule is visible on ultrasound without significant extension posterior to trachea or mediastinal component
* Selected nodule is amenable to trans-isthmus approach
* Normal complete blood count, blood coagulation, serum levels of thyroid hormones, thyrotropin (TSH), calcitonin, and absence of anti-thyroglobulin antibodies (TgAb) and anti-thyroid peroxidase antibodies (TPOAb)
* Patient agrees to participate in the clinical study and to complete all required visits and evaluations
* Negative serum or urine pregnancy test for females of childbearing potential at base line pre-procedure evaluation

Exclusion Criteria:

* Patients with cardiac arrhythmia and/or implanted cardiac device
* Hyper-functioning nodules, evaluated by thyroid function test and/or 99mTc-pertechnetate scintigraphic findings
* History of neck radiation therapy
* Pregnancy
* Allergies to medications for anesthesia
* Primary thyroid PTC with aggressive histology (tall cell, columnar cell, insular, e.g.) in consultation with cytology, endocrine and surgery team
* Extra-thyroidal invasion of PTC OR local nodal/distant systemic metastatic disease
* Cystic nodules (< 70% solid components)
* Calcified nodules
* Targeted nodule within 0.5 cm from the major vessels, vagus nerve, brachial plexus, and recurrent laryngeal nerve
* Patients with contralateral vocal cord paralysis
* Uncorrectable coagulopathy with partial thromboplastin time (PTT) > 1.5 x upper limit of normal (ULN) or international normalized ratio (INR) > 1.5 or platelet count <100,000 per mm^3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Changes in thyroid nodule size | Baseline up to 12 months
  The change from baseline to follow-up will be evaluated using Wilcoxon signed-rank tests. Additionally, will assess the association between changes in the nodule volume and covariates of interest, including but not excluded to the percentage of volume ablated, the nodule composition at treatment and follow-up, and the amount of energy delivered in Joules.

SECONDARY OUTCOMES:
Treatment response that affect quality of life | Up to 12 months post-treatment
  Will compare symptom scores and cosmetic grades to baseline using Wilcoxon signed-rank tests at both 6 months and at 12 months of follow-up.
Sonographic features of nodules | Up to 12 months post-treatment
  Sonographic features will be summarized descriptively.
Cost of ultrasound-guided radiofrequency ablation (RFA) | Up to 12 months post-treatment
  The cost of ultrasound-guided RFA will be summarized. Comparisons may be made with historical data on the costs associated with surgical thyroidectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Kim O Learned, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT05003856/ICF_000.pdf